CLINICAL TRIAL: NCT01347372
Title: Peer to Peer Mentoring For Individuals With Early Inflammatory Arthritis: An Effectiveness Study (Pilot RCT)- Peer Mentor Training
Acronym: P2P EIA RCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sunnybrook Health Sciences Centre (Other)
Collaborators: Canadian Rheumatology Association (Other); The Arthritis Society, Canada (Other); Mount Sinai Hospital, Canada (Other); Unity Health Toronto (Other); University of Toronto (Other)
Responsible Party: Principal Investigator, Dr. Mary Bell, Rheumatologist, Sunnybrook Health Sciences Centre
Allocation: Not Applicable | Model: Single Group | Purpose: Health Services Research
Other Study IDs: 095-2011
Record Dates: First submitted 2011-05-02; First posted 2011-05-04 (Estimated); Last update posted 2018-04-12 (Actual); Status verified 2018-04

CONDITIONS: Early Inflammatory Arthritis
Keywords: peer support; peer mentoring; peer counselling; arthritis; chronic disease; inflammatory arthritis; early inflammatory arthritis; rheumatoid arthritis
MeSH Terms: conditions — Arthritis; Chronic Disease; Arthritis, Rheumatoid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: Peer Mentor Training — Peer mentors will complete a training program (up to 20 hours) during which they will be evaluated. This face-to-face training applies an interactive format, with a combination of lectures, question/answer sessions, and experiential learning (e.g. role-playing, simulations) and practice sessions.

SUMMARY:
Peer support (including informational, emotional, appraisal support) has been shown to help persons with chronic conditions. The goal of this research is to examine the impact of early peer support on the health and quality of life of individuals with early inflammatory arthritis (EIA). The investigators hypothesize that early peer support will result in improved use of disease modifying anti-rheumatic drug (DMARD) or biologic treatment, self-efficacy, coping efficacy, social support, health-related quality of life, self-management, and disease activity score as well as reduced anxiety for individuals with EIA within 2 years of their diagnosis. In this study, persons with IA will be trained as peer mentors using a training program developed for a pilot study. Individuals with EIA will be randomized to receive either "peer support program" or "standard care". Peer mentors will be paired with a person with EIA to provide one-on-one support (face-to-face or telephone) once a week for approximately 30 minutes over a 12-week period. All "standard care" participants will receive the peer mentoring intervention at the end of study. Both groups will be evaluated using self-administered questionnaires and clinical assessments, and results of the two groups will be compared. This information will be used to design a larger study.

DETAILED DESCRIPTION:
Background: The investigators are proposing to examine the effectiveness of a peer support program, the aim of which is to assist individuals with early inflammatory arthritis (EIA) to receive the education and support they need to make decisions to manage their disease. Peer support (including informational, emotional, appraisal support) has been shown to assist persons with chronic conditions and may address challenges with receiving timely and proper treatment in persons with EIA.

Purpose: The goal of this pilot randomized controlled trial (RCT) is to evaluate the effectiveness of peer support to improve the health and quality of life of individuals with EIA. The investigators hypothesize that early peer support will result in improved use of treatment, self-efficacy, coping efficacy, social support, health-related quality of life, self-management, and disease activity score, as well as reduced anxiety for individuals with EIA within two years of their diagnosis.

Methods: This proposal builds on a pilot study, currently underway, to develop and evaluate the acceptability and feasibility of a peer support intervention for persons with EIA. The proposed effectiveness study will employ a RCT design with a wait list control group. Individuals with IA (diagnosis 2 or more years) will be trained as peer mentors using the revised pilot study training program. Peer mentors will be matched with a person newly diagnosed with IA to provide one-on-one support (face-to-face or telephone) over a 12-week period. Individuals with EIA will be recruited from rheumatology clinics at Sunnybrook Health Sciences Centre and Mount Sinai Hospital. Individuals with EIA will be randomized to either "intervention" or "standard care" (wait list). All "standard care" participants with EIA will receive the peer mentoring program at the end of study period; their outcomes will be also be evaluated. Both "intervention" and "standard care" participants will complete clinical assessments and self-administered questionnaires before and after (immediate post-program and 3-month follow-up) study completion to evaluate use of treatment, self-efficacy, coping efficacy, social support, health-related quality of life, anxiety, self-management, and disease activity count.

Implication: The study aims to improve the education and support for patients with EIA. The data from this study will be used to further refine the intervention and study design to be subsequently submitted for further effectiveness testing in a larger scale RCT.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of IA from a physician;
* Disease duration at least 2 years and managing well;
* Currently using medications (DMARDS/biologics) to treat his/her arthritis
* Completion of Arthritis Self-Management Program (ASMP) provided by The Arthritis Society and/or similar program and/or have sufficient knowledge and experience with teaching or providing mentoring support to an individual living with a chronic disease;
* Able to attend a series of training sessions (approximately 20 hours in total);
* Able to take part in ongoing assessment/evaluation activities (self-report questionnaire; interviews, observation; study activity log)
* Able to commit to the duration of the research study (9 -12 months);
* Willing to provide ongoing one-on-one support to an individual newly diagnosed with IA;
* 18 years of age or older; and
* Able to speak, understand, read and write English.

Exclusion Criteria:

•

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2011-05 (Actual); Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
self-efficacy | 0 months (baseline); immediate post-training; immediate post peer mentoring intervention and 3 months follow-up post peer mentoring intervention
  The primary goals of this study are to increase peer mentors' knowledge, confidence, skills and abilities to provide one-on-one support to individuals with EIA. It is anticipated that after training, peer mentors will be able to provide support to help persons with EIA to make informed decisions to self-manage their disease.

CONTACTS AND LOCATIONS:
Overall Officials: Mary J Bell, MD, FRCPC, Principal Investigator — Sunnybrook Health Sciences Centre
Locations (2):
- Canada (2):
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
  - Mount Sinai Hospital, Toronto, Ontario